CLINICAL TRIAL: NCT03433352
Title: The Effect of Intestinal Microbiota on Treatment Sensitivity and Prognosis of Methimazole for GD
Brief Title: Intestinal Microbiota and Treatment of GD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2017-12-23
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2017-12

CONDITIONS: Microbiota
Keywords: gut microbiota; 16S rRNA gene; Graves' disease; Methimazole; Propylthiouracil
MeSH Terms: conditions — Graves Disease | interventions — Methimazole; Propylthiouracil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control group: 30 healthy volunteers were included in the healthy control group
- Recrudescence group: 30 GD patients who received recurrence within 2 years after treatment with Methimazole Pill or propylthiouracil pill
  Interventions: Drug: Methimazole Pill; Drug: Propylthiouracil Pill
- No recrudescence group: 30 GD patients who did not receive recurrence within 2 years after treatment with Methimazole Pill or propylthiouracil pill
  Interventions: Drug: Methimazole Pill; Drug: Propylthiouracil Pill

INTERVENTIONS:
Drug: Methimazole Pill — Patients who developed GD received methimazole treatment
  Groups: No recrudescence group; Recrudescence group
Drug: Propylthiouracil Pill — Patients who developed GD received propylthiouracil treatment
  Groups: No recrudescence group; Recrudescence group

SUMMARY:
Graves' disease is an organ-specific autoimmune disease in which both genetic predisposition and environmental factors serve as disease triggers. Many studies have indicated that alterations in the gut microbiota are important environmental factors in the development of inflammatory and autoimmune diseases. Investigators systematically performed a comparative analysis of the gut microbiota in GD patients and healthy controls and analyse the relationship between intestinal microbiota and GD drug therapy.

DETAILED DESCRIPTION:
Graves' disease is an organ-specific autoimmune disease in which both genetic predisposition and environmental factors serve as disease triggers. Many studies have indicated that alterations in the gut microbiota are important environmental factors in the development of inflammatory and autoimmune diseases. Investigators systematically performed a comparative analysis of the gut microbiota in GD patients and healthy controls before and found that gut microbiota changed between GD patients and healthy controls.But there are few articles on the relationship between intestinal microbiota and drug treatment of GD, so Investigators explored the relationship between intestinal microflora and methimazole treatment for GD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* GD was clinical diagnosed and accept the standard treatment of methimazole or propylthiouracil and thyroid function returned to normal

Exclusion Criteria:

* Pregnancy
* Lactation
* Cigarette smoking
* Alcohol addiction
* Hypertension
* Diabetes mellitus
* Lipid dysregulation
* BMI > 27
* Recent (< 3 months prior) use of antibiotics, probiotics, prebiotics, symbiotics, hormonal medication, laxatives, proton pump inhibitors, insulin sensitizers or Chinese herbal medicine
* History of disease with an autoimmune component, such as MS, rheumatoid arthritis, IBS, or IBD
* History of malignancy or any gastrointestinal tract surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients were included according to the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-12-23 (Actual); Primary Completion 2018-12-23 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Transcriptional changes in gut microbiota | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months and 24 month respectively after Methimazole withdrawal
  The microbiota measured by 16S rRNA gene

SECONDARY OUTCOMES:
Serum thyroid function changed | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months and 24 month respectively after Methimazole withdrawal
  Serum thyroid function measured by Immunohistochemistry

OTHER OUTCOMES:
Serum thyroid related antibodies changed | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months and 24 month respectively after Methimazole withdrawal
  Serum thyroid related antibodies measured by Immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Yunwei Wei, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calissendorff J, Mikulski E, Larsen EH, Moller M. A Prospective Investigation of Graves' Disease and Selenium: Thyroid Hormones, Auto-Antibodies and Self-Rated Symptoms. Eur Thyroid J. 2015 Jun;4(2):93-8. doi: 10.1159/000381768. Epub 2015 May 27. PMID 26279994
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967